CLINICAL TRIAL: NCT07198997
Title: Comparison of the Effects of Intraosseous Anesthesia Performed With the SleeperOne5 Computer-Controlled Device and Conventional Mandibular Nerve Block on Behavior and Pain Control During Anesthesia Administration in Children Aged 5-9: A Randomized Clinical Trial
Brief Title: Comparison of the Effects of Intraosseous Anesthesia Performed With the SleeperOne5 Computer-Controlled Device and Conventional Mandibular Nerve Block on Behavior and Pain Control During Anesthesia Administration in Children Aged 5-9
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Pelin Turan, PhD student, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: SPZ001
Record Dates: First submitted 2025-07-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: the Impact of Modern Anesthesia Techniques Applied in Pediatric Dentistry on Physiological Parameters
Keywords: anxiety reduction, CCLA, digital anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital intraosseous anesthesia (Experimental)
  Interventions: Other: digital anesthesia
- conventional mandibular nerve block anesthesia. (Active Comparator)
  Interventions: Other: digital anesthesia

INTERVENTIONS:
Other: digital anesthesia — mandibular anestezi ile digital intrsosseoz anesteziyi kıyasslayan calısma yok.

SUMMARY:
The injection stage is the most intense cause of anxiety during dental treatment in the pediatric patient group. It is aimed to keep the pain sensation at a minimum during this process. Computer-controlled local anesthesia delivery systems that can inject anesthetic solution at a fixed rate, pressure and volume have been developed in order to reduce pain, discomfort, anxiety and control the injection flow. This study aimed to compare the behavioral and physiological differences in children between the computer-controlled intraosseous anesthesia technique and conventional inferior alveolar nerve blockade. 100 systemically healthy children aged 6-9 years with contralateral pulpotomy or pulpectomy of the mandible and the 2nd primary molar tooth will be included in this study. During the application of local anesthesia, heart rate, which is a physiological criterion, will be measured in the assessment of pain. For this purpose, fingertip pulse oximeter will be used. The child's cooperation level during the treatment process will be evaluated using the Venham behavioral rating scale. The "visual analog scale" will be shared with the patients and the pain perception during the treatment process will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* One hundred systemically healthy children aged 6 to 9 years, with Frankl Behavior Scale scores of 3 and 4, who have not used any analgesics within 48 hours prior to the study.

Exclusion Criteria:

* Children with teeth exhibiting mobility, necrosis, furcation involvement, or periapical radiolucency, and children who do not have contralateral second primary molars in different quadrants of the mandible.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Pain and behavioral response during local anesthesia administration, heart rate, venham behavior rating scale | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: ŞÜKRİYE T KAYACI, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)